CLINICAL TRIAL: NCT01454791
Title: Diclofenac Sodium Topical Gel to Reduce Injection Site Discomfort in Patients With Multiple Sclerosis Taking Glatiramer Acetate: A Randomized Controlled Double- Blind Crossover Trial
Brief Title: Diclofenac Sodium Topical Gel to Reduce Injection Site Discomfort in Patients Taking Glatiramer Acetate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brown, Theodore R., M.D., MPH (Individual)
Collaborators: Teva Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: WIRB 20101775
Record Dates: First submitted 2011-08-09; First posted 2011-10-19 (Estimated); Results first posted 2015-02-13 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; diclofenac; subcutaneous injection; glatiramer acetate; Copaxone
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac Sodium Topical Gel first then Placebo (Experimental): 1:1 randomization to either of two treatment phases of 2 weeks duration (active-placebo or placebo-active).
  Interventions: Drug: diclofenac sodium topical gel; Other: Placebo
- Placebo first then Diclofenac Sodium Topical Gel (Placebo Comparator): 1:1 randomization to either of two treatment phases of 2 weeks duration (active-placebo or placebo-active).
  Interventions: Drug: diclofenac sodium topical gel; Other: Placebo

INTERVENTIONS:
Drug: diclofenac sodium topical gel — diclofenac sodium topical gel 1% applied 1-4 times per day for two weeks either preceded by or followed by two weeks of placebo
  Other Names: Voltaren gel
Other: Placebo — a placebo gel is applied 1-4 times per day for two weeks.

SUMMARY:
The purpose of this study is to assess the effect of Diclofenac Sodium Topical Gel (DSTG) on injection site reaction following self-administer glatiramer acetate in people with Multiple Sclerosis.

DETAILED DESCRIPTION:
A 4 week study with active or placebo medication at randomization and switch treatment at 2-week crossover visit (2 weeks on each arm). There will be a total of 3 visits to the clinic. Subjects will receive instruction on how to apply the DSTG/placebo at the injection site and keep a daily injection site reaction diary.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis (MS) made at least 3 months prior based on McDonald or Poser criteria.
* Age 18 or more
* Ongoing treatment with glatiramer acetate (Copaxone) for three months or more.
* No MS exacerbation for 60 days prior to screening.
* Mean score of greater than or equal to 1.0 on screening Local Injection Site Reaction scale of last 3 days.
* Written informed consent.

Exclusion Criteria:

* Regular use of any non-steroidal anti-inflammatory drug (NDAID), except Asprin (<325 mg daily), between screening and end of study.
* Any contraindication to Diclofenac Sodium Topical Gel (DSTG)

  * allergy to DSTG or any NSAID.
  * history of asthma, urticaria, or other allergic reaction after taking any NSAID.
* Females who are breast feeding, pregnant or have potential to become pregnant during the course of the study(fertile and unwilling/unable to use effective contraceptive measures).
* Cognitive deficits that would interfere with the subject's ability to give informed consent or preform study testing.
* Any other serious and/or unstable medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ted R Brown, MD, MPH, Principal Investigator — MS Center at Evergreen Healthcare
Locations (1):
- MS Center at Evergreen Healthcare, Kirkland, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Diclofenac Sodium Topical Gel Followed by Placebo: diclofenac sodium topical gel: diclofenac sodium topical gel 1% applied 1-4 times per day for two weeks followed by two weeks of placebo
  Placebo: a placebo gel is applied 1-4 times per day for two weeks.
- Placebo Followed by Diclofenac Sodium Topical Gel: Placebo for two weeks followed by diclofenac sodium topical gel: diclofenac sodium topical gel 1% applied 1-4 times per day for two weeks
  Placebo: a placebo gel is applied 1-4 times per day for two weeks.
Period: Overall Study
Arm/Group | Diclofenac Sodium Topical Gel Followed by Placebo | Placebo Followed by Diclofenac Sodium Topical Gel
Started | 20 | 20
Completed | 20 (20 subjects started with Diclofenac, then switched to placebo) | 20 (20 subjects started with placebo, then switched to Diclofenac)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Followed by Diclofenac Sodium Gel: placebo for 2 weeks followed by diclofenac sodium topical gel: diclofenac sodium topical gel 1% applied 1-4 times per day for two weeks
  Placebo: a placebo gel is applied 1-4 times per day for two weeks.
- Total: Total of all reporting groups
Arm/Group | Diclofenac Sodium Topical Gel Followed by Placebo | Placebo Followed by Diclofenac Sodium Gel | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Local Injection Site Reaction (0-6) Scale at Baseline, 2 Weeks
Description: patients will complete a daily diary rating their reaction for elements including pain and inflammation or no reaction to all 6 elements listed on the local injection site reaction scale. Range of scores is 0-6 with zero best and 6 worst.
Time Frame: 2 weeks
Population: The primary outcome is looking at between-intervention differences at 2 weeks of intervention. Not a comparison at any other timepoint
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Diclofenac Sodium Topical Gel: diclofenac sodium topical gel: diclofenac sodium topical gel 1% applied 1-4 times per day for two weeks
- Placebo: Placebo for 2 weeks: a placebo gel is applied 1-4 times per day.
Arm/Group | Diclofenac Sodium Topical Gel | Placebo
Number analyzed (Participants) | 40 | 40
units on a scale | 3.39 (0.19) | 3.47 (0.19)
Statistical Analysis 1: Comparison: Diclofenac Sodium Topical Gel vs Placebo; Test type: Superiority or Other; p = 0.45, t-test, 2 sided; Mean Difference (Final Values) = -0.08

2. Primary Outcome: Pain Scale at 2 Weeks
Description: 0-10 subjective Likert scale for severity of injection site reaction associated pain. Zero is best and 10 is worst
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diclofenac Sodium Topical Gel | Placebo
Number analyzed (Participants) | 40 | 40
units on a scale | 2.44 (0.28) | 2.60 (0.28)
Statistical Analysis 1: Comparison: Diclofenac Sodium Topical Gel vs Placebo; Test type: Superiority or Other; p = 0.6059, t-test, 2 sided; Mean Difference (Final Values) = -0.16 — not significant

3. Secondary Outcome: Subject Global Impression at 2 Weeks
Description: This is a single question: "How would you rate your level of comfort with Copaxone injection during the past two weeks?" Responses include Extremely good, Quite good, Better than average, Average, Below Average, Quite bad, Extremely bad.
Time Frame: 2 weeks
Population: The secondary outcome is looking at between-intervention differences at 2 weeks of intervention. Not a comparison at any other timepoint
Measure: Mean (Standard Deviation); unit: Likert scale 1-7 (7= best)
Groups:
- Placebo: Placebo for two weeks: a placebo gel is applied 1-4 times per day
Arm/Group | Diclofenac Sodium Topical Gel | Placebo
Number analyzed (Participants) | 40 | 40
Likert scale 1-7 (7= best) | 4.68 (0.17) | 4.50 (0.17)
Statistical Analysis 1: Comparison: Diclofenac Sodium Topical Gel vs Placebo; Test type: Superiority or Other; p = 0.705, t-test, 2 sided; Mean Difference (Final Values) = 0.18 — not significant

ADVERSE EVENTS:
Groups:
- Diclofenac Sodium Topical Gel; Placebo: 1:1 randomization to either of two treatment phases of 2 weeks duration (active-placebo or placebo-active).
  diclofenac sodium topical gel: diclofenac sodium topical gel 1% applied 1-4 times per day for two weeks either preceded by or followed by two weeks of placebo
  Placebo: a placebo gel is applied 1-4 times per day for two weeks.
Arm/Group | Diclofenac Sodium Topical Gel | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Sodium Topical Gel (N=20) | Placebo (N=20)
urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No